CLINICAL TRIAL: NCT02304653
Title: Acute Appendicitis: The Influence of C-reactive Protein and Leucocytes on Clinical Decision-making
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Niels Qvist, Professor, Odense University Hospital
Other Study IDs: 12-132020
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Clinical descision making — Chage in diagnosis before and after the presentation of the reults of CRP and Leucocytes

SUMMARY:
Aim: To investigate if the results of CRP and leucocytes had any positive or negative influence on the surgeon's decision-making when handling patients with suspected AA.

DETAILED DESCRIPTION:
A prospective observational cohort study including patients (≥15 years of age) admitted on suspicion of AA. The surgeons were instructed to perform their physical examination and register whether they found the patient more or less than 50% likely to have AA. Thereafter, the surgeons had to assess the blood results and reevaluate their diagnosis. The surgeon's diagnosis before and after was compared to the final diagnosis defined by surgical findings or follow up. Gold standard was any degree of appendicitis on histology.

ELIGIBILITY:
Acutae abdominal pain Suspect for acute appendicites

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute abdominal pain with the suspicion of acute appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in diagnosis | Two hours

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Study Director — Head of surgical eserach unit
Locations (1):
- Odense University Hospital, surgical department A, Odense C, Denmark

REFERENCES:
- [Derived] Tind S, Qvist N. Acute Appendicitis: A Weak Concordance Between Perioperative Diagnosis, Pathology and Peritoneal Fluid Cultivation. World J Surg. 2017 Jan;41(1):70-74. doi: 10.1007/s00268-016-3686-8. PMID 27541029
- [Derived] Tind S, Lassen AT, Zimmerman-Nielsen E, Qvist N. C-reactive protein and white blood cell count do not improve clinical decision-making in acute appendicitis. Dan Med J. 2015 Dec;62(12):A5167. PMID 26621395